CLINICAL TRIAL: NCT05272033
Title: The Effect of Transcutaneous Electrical Acupoint Stimulation (TEAS) on Prevention Hypotension Related to Spinal Anesthesia in Elderly Patients
Brief Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) on Prevention Hypotension in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TEAS Elderly Hypotension
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP TEAS (Active Comparator): Patients in the TEAS group will receive preoperative TEAS for 30 min before the spinal anesthesia at PC-5, PC-6, and ST-36 with an electronic acupuncture device.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation
- Sham TEAS (Sham Comparator): In the sham TEAS group, the gel electrodes will be applied at the same anatomical points without stimulation.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Acupoint Stimulation — Transcutaneous Electrical Acupoint Stimulation

SUMMARY:
Despite prophylactic measures, hypotension remains a common side-effect of spinal anesthesia. Electroacupuncture influences hemodynamics. We hypothesized that transcutaneous electrical acupuncture point stimulation (TEAS) at traditionally used acupuncture points would reduce the severity of hypotension after spinal anesthesia in geriatric patients undergoing hernia surgery.

DETAILED DESCRIPTION:
After obtaining written informed patient consent, 60 geriatric patients undergoing hernia surgery under spinal anesthesia were randomized into two groups. In the placebo TEAS group, the gel electrodes will be applied at the same anatomical points without stimulation. The acupoint group will receive TEAS at the PC-5, PC-6, and ST-36 points bilaterally before the spinal anesthesia. The spinal anesthesia will be performed using 12.5 mg 0.5% bupivacaine was from the L3-4 or L4-5 interval with a 25G Quincke spinal needle. Hemodynamic data will be followed every five minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients aged 65 years and older who are scheduled for inguinal hernia repair

Exclusion Criteria:

* Patients with neurological or psychological diseases
* Patients who have been treated with TEAS or acupuncture before,
* Patients with heart failure and pace-maker
* Those who have a local infection in the TEAS area.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
patients blood pressure will be measured | 30 minutes following spinal anesthesia
  Hypotension was defined as a preoperative systolic measurement of >20% or a systolic blood pressure below 100 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)